CLINICAL TRIAL: NCT04236440
Title: Proof-of-mechanism Single-center, Randomized, Double-blind, Placebo-controlled 2-way Crossover Study to Investigate Pharmacodynamics, Safety, Tolerability and Exposure of BAY 2586116 (Part A) and an Open-label Comparison of Different Application Modes for Single Nasal/Pharyngeal Dose Administrations (Part B and Part C) in 12 Participants With Obstructive Sleep Apnea
Brief Title: Study on the Safety of Drug BAY2586116 and How it Works in Patients With Obstructive Sleep Apnea (a Sleep Disorder Caused by the Narrowing and Collapse of the Airway During Sleep) Including the Blood Level of the Drug and Effect of Its Doses and Routes of Administration
Acronym: KOALA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20732
Record Dates: First submitted 2020-01-21; First posted 2020-01-22 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — L 644711

STUDY DESIGN:
Intervention Model Description: Part A: placebo-controlled 2-way crossover Part B: fixed single sequence Part C: single group, single dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A: Randomized, double-blind Part B: Open-label Part C: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: A1A2+Part B+Part C (Experimental): Part A: Participants will receive a single dose administration of BAY2586116 (A1) in treatment period 1, and a single dose administration of placebo (A2) in treatment period 2.
  Part B: After successfully completing Part A, participants will proceed to Part B of the study.
  Participants will receive a single dose administration of BAY2586116 (B1) in treatment period 3.
  Based on the result of the interim analysis there are two possible scenarios regarding mode of application and doses of BAY2586116 to be administered in treatment period 4: 1) a single dose administration of BAY2586116 (B2) Or 2) a single dose administration of BAY2586116 (B3).
  Part C: Participants completing Part B will be invited to participate in an additional treatment period with a single dose BAY2586116 (C).
  Interventions: Drug: BAY2586116 (A1); Drug: Placebo (A2); Drug: BAY2586116 (B1); Drug: BAY2586116 (B2); Drug: BAY2586116 (B3); Drug: BAY2586116 (C)
- Part A: A2A1+Part B+Part C (Experimental): Part A: Participants will receive a single dose administration of placebo (A2) in treatment period 1, and a single dose administration of BAY2586116 (A1) in treatment period 2.
  Part B: After successfully completing Part A, participants will proceed to Part B of the study.
  Participants will receive a single dose administration of BAY2586116 (B1) in treatment period 3.
  Based on the result of the interim analysis there are two possible scenarios regarding mode of application and doses of BAY2586116 to be administered in treatment period 4: 1) a single dose administration of BAY2586116 (B2) Or 2) a single dose administration of BAY2586116 (B3).
  Part C: Participants completing Part B will be invited to participate in an additional treatment period with a single dose BAY2586116 (C).
  Interventions: Drug: BAY2586116 (A1); Drug: Placebo (A2); Drug: BAY2586116 (B1); Drug: BAY2586116 (B2); Drug: BAY2586116 (B3); Drug: BAY2586116 (C)

INTERVENTIONS:
Drug: BAY2586116 (A1) — 160 μg BAY2586116 (nasal spray administration)
Drug: Placebo (A2) — Placebo matching BAY2586116 (nasal spray administration)
Drug: BAY2586116 (B1) — 160 μg BAY2586116 (nasal drops)
Drug: BAY2586116 (B2) — 80 μg BAY2586116 (nasal spray)
Drug: BAY2586116 (B3) — 160 μg BAY2586116 (pharyngeal spray with direct endoscopic application via a nostril)
Drug: BAY2586116 (C) — 160 μg BAY2586116 (pharyngeal spray with direct endoscopic application via a nostril). It is the same procedure as described under part B3.

SUMMARY:
The researchers in this study want to learn how drug BAY2586116 works in patients with obstructive sleep apnea (OSA). OSA is a sleep disorder marked by breathing pauses during sleep due to repetitive obstructions of the upper airway. BAY2586116 is a new drug under development for the treatment of OSA. It blocks protein channels expressed on the surface of the upper airways in small mechanoreceptors (a type of molecule that sense and pass stimulus outside a cell on to the inside of the cell through mechanical gate on the surface of the cell). Thus, the negative pressure reflex alerting the brain of inspiration is triggered more easily leading to a stronger activation of throat muscles. This prevents narrowing or collapse of the upper airways during sleep which is one of the pathological key factors in OSA.

Researchers will study the effects of different routes of administration (drops into the nose, spray into the nose or throat or spray into the throat by endoscopy). Endoscopy allows the doctor to look at areas in the throat that cannot be seen with a mirror: a thin tube-like instrument is inserted through the nose to check and give the medication. Different doses of the test drug will be given.

They also want to find out if participants experience any medical problems during the study.

Patients participating in this study will undergo three study parts. After completing Part A and Part B, participants will be asked to join Part C. In Part A, participants will receive both the test drug and placebo (a placebo looks like the test drug but does not have any medicine in it); in Part B, participants will receive the test drug twice via different routes of administration (drops in nose and spray in nose or throat) and in Part C, the participants would receive the test drug once via spray in throat by endoscopy. The sleep of the participants will be monitored by medical equipment. Participants will be asked to visit the clinic 7 times in 14 weeks in total.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age or above at the time of signing the informed consent.
* Participants need to be diagnosed with OSA but should be considered otherwise healthy at the discretion of the investigator.
* Participants do not need to be on CPAP therapy at the time of the study. However, if they are on therapy, participants must commit to keep their treatment schedule constant during the study period, especially the night before each administration of study intervention. For participants on CPAP, this will be monitored objectively using the compliance chip within the CPAP devices.
* Female of non-child bearing potential or male.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  1. Female participants:

     -- i. Participants of non-childbearing potential, i.e. post-menopausal (no menses for at least 1 year) or surgically sterile (documented history of tubal ligation, hysterectomy or bilateral oophorectomy).
  2. Male participants:

     * i. Male participants of reproductive potential must agree to utilize two reliable and acceptable methods of contraception simultaneously when sexually active. This applies for the time period between admission to the study site until 12 weeks after the last administration of the study intervention.

Acceptable methods of contraception include, but are not limited to, (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Ability to understand and follow study-related instructions.
* The informed consent must be signed before any study specific tests or procedures are done. For Part C reconsent must be signed.

Exclusion Criteria:

* Severely impaired breathing within two days prior to randomization (e.g. acute nasal congestion during upper airway infection).
* Subject with known allergies or hypersensitivities to the study drugs (active substances or excipients of the preparations).
* Any other condition which at the discretion of the investigator would make the participant unsuitable for participation in the study and will not allow participation for the full planned study period (e.g. active malignancy or other condition limiting life expectancy to less than 12 months).
* Use of any topical medication containing local anesthetics for nose and throat within 2 days before each administration of study intervention.
* Donation of more than 100 mL of plasma or equivalent volume of blood within 4 weeks or 500 mL whole blood within 3 months before study drug administration.
* Previous participation in this study.
* Participation in another clinical study with study intervention(s) within 90 days prior to first administration.
* Heavy smoking, i.e. more than 20 cigarettes per day.
* Light smokers who are unable to cease smoking for the duration of the inhouse phases of the study (i.e. Study day 1 in treatment periods 1, 2, 3 and 4).
* Drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Critical closing pressure (Pcritgs) of the upper airway (cmH2O) during sleep with a polysomnography | From start of sleep to end of sleep of administration day (Day 1)

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From first application of study intervention up to 2 days after end of treatment with study intervention in each period
Severity of treatment-emergent adverse events (TEAEs) | From first application of study intervention up to 2 days after end of treatment with study intervention in each period

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaide Institute for Sleep Health, Bedford Park, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be later determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Osman AM, Mukherjee S, Altree TJ, Delbeck M, Gehring D, Hahn M, Lang T, Xing C, Muller T, Weimann G, Eckert DJ. Topical Potassium Channel Blockage Improves Pharyngeal Collapsibility: A Translational, Placebo-Controlled Trial. Chest. 2023 Apr;163(4):953-965. doi: 10.1016/j.chest.2022.11.024. Epub 2022 Nov 24. PMID 36435266
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/